CLINICAL TRIAL: NCT05399043
Title: Perception of High Technology in Rehabilitation: a Prospective Real-life Study on Usability, Effectiveness, and Health-related Quality of Life (PHTinRehab Study)
Brief Title: Experience of Use and Biopsychosocial Effects of Robotic and Virtual Reality Devices in Neuromotor Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Antonia Pierobon, Psychologist, Istituti Clinici Scientifici Maugeri SpA
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2517
Record Dates: First submitted 2022-04-22; First posted 2022-06-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2023-09

CONDITIONS: Neurologic Diseases; Arthropathy of Knee; Arthropathy of Hip
Keywords: Acquired Brain Injury; Parkinson's Disease; Total Knee Arthroplasty; Total Hip Arthroplasty; Robot-Assisted Therapy; Virtual Reality; Health-related Quality of Life; Cognitive Functioning; Usability
MeSH Terms: conditions — Nervous System Diseases; Brain Injuries; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel, non-randomized prospective quasi-experimental study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Technology-based Rehabilitation Group (Experimental): Patients will undergo conventional treatment and, additionally, robot-assisted therapy or virtual reality-based rehabilitation.
  Interventions: Other: Multidisciplinary Conventional Neuromotor Rehabilitation; Device: Technology-based Rehabilitation
- Conventional Rehabilitation Group (Active Comparator): Patients will undergo conventional treatment exclusively.
  Interventions: Other: Multidisciplinary Conventional Neuromotor Rehabilitation

INTERVENTIONS:
Other: Multidisciplinary Conventional Neuromotor Rehabilitation — Patients will receive conventional treatment consisting of two daily one-hour session (4 weeks) and including traditional rehabilitation activities like range of motion exercises (passive, active assisted and active), progressive resistive exercises, balance and strength training, and aerobic conditioning. The intervention procedures will follow the routine multidisciplinary clinical practice of the Institute where the study will be carried out. Procedures will be adapted according to patient's medical diagnosis, disability severity, and to the consequent rehabilitation objectives in favor of an individualized rehabilitation project and program. If necessary, patients might therefore undergo parallel rehabilitation activities (ie, occupational therapy, speech therapy, cognitive stimulation) that will be kept under control throughout data collection and analyses.
Device: Technology-based Rehabilitation — According to their individualized rehabilitation project, patients will undergo RAT or non-immersive VR-based rehabilitation.
  RAT will consist of three times a week one-hour session (4 weeks) and will be conducted by the implementation of an exoskeleton device for the upper limbs (Armeo-Spring™) or for the lower limbs (Lokomat™).
  VR-based rehabilitation will consist of one daily one-hour session (4 weeks) and will be conducted by the implementation of a single non-immersive VR device among the Riablo™ (Corehab, Italy), the ProKin 252™ (TechnoBody SRL, Italy), the D-Wall™ (TechnoBody SRL, Italy), the Walker View™ (TechnoBody SRL, Italy).
  Part of the duration of the whole treatment will be dedicated to the use of the device, resulting in the same amount of rehabilitation for all participants.
  Arms: Technology-based Rehabilitation Group

SUMMARY:
The implementation of virtual reality (VR) and robotic devices in neuromotor rehabilitation has so far provided promising evidence in terms of efficacy throughout different clinical populations. Positive changes in patient's motor and functional outcomes were reported along with an increased autonomy in the activities of daily living (ADLs) and health-related quality of life (HRQoL). The experience of use of these technological devices and their impact on the cognitive and psychosocial outcomes remain still unclear, though. Adopting a biopsychosocial approach, the present two-arm, parallel, non-randomized prospective quasi-experimental study protocol aims to explore the short- and long-term effectiveness of robot-assisted therapy (RAT) and of VR-based neuromotor rehabilitation. Pre-post intervention effects will be estimated and compared between a group of patients undergoing conventional treatment and another group additionally participating in technology-based rehabilitation. The evaluation will include patient's functional status (ie, motor functionality, autonomy in ADLs, risk of falls), cognitive functioning (ie, attention and executive functions), HRQoL, and psychological aspects (ie, anxiety and depression symptoms, quality of life satisfaction). After the treatment, devices usability and experience of use, along with the related psychosocial impact will be also assessed.

DETAILED DESCRIPTION:
Over the past two decades, the aging population and the related increase of acute and chronic diseases have led to the need for urgent healthcare solutions, including the implementation of interdisciplinary and innovative approaches in patients' care. Contextually, the field of neuromotor rehabilitation has shown deep interest in the deployment of robotic and virtual reality (VR) devices in recovery programs, given their multipurpose application.

Robot-assisted therapy (RAT) has reported promising evidence so far, showing advantages like the possibility to provide repetitive, intensive, and task-oriented rehabilitation activities, including the opportunity to implement smaller workforce, optimized exercise, and real-time quantitative motor assessment and monitoring. To date, diverse robot typologies (ie, exoskeletons, end-effectors, soft-robots) have been implemented to treat different chronic and complex diseases like acquired brain injury (ABI), spinal cord injury (SCI), multiple sclerosis (MS), and Parkinson's disease (PD) reporting evidence in favor of their feasibility and an improvement in patient functionality, autonomy and health-related quality of life (HRQoL).

Likewise, VR has been shown to be a promising tool to enhance rehabilitation outcomes. When various technical devices (eg, head-mounted displays, motion capture and tracking systems) are implemented, it can deliver realistic experiences by interacting with virtual environments (VEs) closely resembling everyday environments. To date, plenty of studies have tested and demonstrated the efficacy, for example, of VR-treadmill trainings for lower limbs, to improve gait and balance, ultimately reducing risk of falls, or of exercises in reaching and grasping virtual objects to target arms and manual movement, dexterity, and coordination. Besides, thanks to the multimodal and multisensory stimulation it can provides, VR has revealed to be an effective tool to obtain significant changes in cognitive outcomes (eg, memory, visual attention, executive functions). Lastly, such stimulation has been shown to have potential for increased patient engagement in the rehabilitation program, ultimately improving treatment compliance.

Nevertheless, alongside the technological devices' complexity and the related clinical application, ensuring adequate patient engagement and adherence to treatment still represents an open challenge. Accordingly, the introduction of technology in rehabilitation programs has raised the issue of devices usability and experience of use. Usability specifically refers to a patient's perception and ability to use a device effectively, efficiently, and satisfactorily. Factors like device ease-of-use and learnability are therefore essential when aiming to achieve adequate technology acceptance rate. Such factors, however, do not always sufficiently explain the complexity of the experience of use. To better expand the concept of device use, socio-cognitive and experiential factors (eg, emotions, motivation, satisfaction) need to be considered too.

In light of the data in the literature, beyond motor and functional recovery what has been scarcely addressed up to date is the potential of RAT and VR to improve patient's psychosocial functioning. Moreover, to optimally enhance technological devices deployment in rehabilitation programs, a deeper understanding on their experience of use is increasingly needed.

Following this line, the purpose of this study protocol is to explore, in a real-world clinical setting, both the experience of use and the biopsychosocial effectiveness of robotic and VR technology in patients undergoing neuromotor rehabilitation. In particular, this protocol outlines the procedures for exploring the perception and the effects of such technology across different neurological (ie, ABI, PD) and orthopedic (ie, total knee/hip arthroplasty) conditions and the implicit differences of the technological devices implemented. Accordingly, within/between-groups observations will be made as appropriate by considering consistent clinical populations and intervention procedures. Specifically, the study objectives are:

1. to explore pre- post-treatment differences and long-term (6-month follow-up) effects concerning: patient's HRQoL, quality of life satisfaction, anxiety and depression symptoms, cognitive functioning, and functional status;
2. to measure patient's perceived experience of the rehabilitation program, as well as the perceived experience of using the robotic and VR devices (user experience and device usability) and the related psychosocial impact;
3. to observe the differences in terms of device experience of use in relation to the pathology, disease severity, and the type of device implemented;
4. to extend the evaluation of the device's perceived usability to the therapists and explore to what extent this is associated to patient's perception of device usability and rehabilitation experience.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Diagnosis of acquired brain injury (ABI) or Parkinson's Disease (PD) or total knee/hip arthroplasty.

Exclusion Criteria:

* severe clinical condition (ie, chronic heart failure [New York Heart Association Classification-IV - NYHA-IV], ischemic heart disease [Canadian Cardiovascular Society Classification-IV - CCS-IV], neoplastic disease, acute respiratory disease);
* severe cognitive impairment (MoCA ≤ 15.5);
* language deficits;
* severe mental health condition or psychiatric disorder compromising participation in the study;
* absence or withdrawal of the informed consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Short-term changes in Modified Barthel Index (MBI) | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The Modified Barthel Index (MBI) evaluates patient's autonomy to perform ADLs (ie, chair/bed transfer, ambulation, stair climbing, toilet transfer, bowel control, bladder control, bathing, dressing, personal hygiene, feeding). Total scores range from 0 to 100. Higher scores indicate higher patient's autonomy.
Short-term changes in Functional Independence Measure (FIM) | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The Functional Independent Measure (FIM) evaluates patient's disability level according to motor and cognitive subscores. Total scores range from 18 (complete dependence) to 126 (complete independence). Two subscores can be calculated: FIM motor (range 13-91) and FIM cognitive (range 5-35).
Short-term changes in Timed Up & Go Test (TUG) | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The Timed Up & Go Test measures patient's risk of falling, static and dynamic balance by estimating the time patient takes to stand up from an armchair, walk forward for 3 meters, turn, walk back to the chair and sit down. The longer the time this takes, the higher the risk of falling.
Short-term changes in Morse Fall Scale (MFS) | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The Morse Falls Scale (MFS) evaluates patient's risk of falls. Total scores ranges from 0 to 125 with higher scores reflecting a greater risk of falling.
Short-term changes in Montreal Cognitive Assessment (MoCA) | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The Montreal Cognitive Assessment (MoCA) test evaluates patient's global cognition (ie, visuospatial abilities, executive functions, attention, concentration, short-term and delayed verbal memory, working memory, language, orientation to time and space). Total scores range from 0 to 30. Higher scores indicate better cognitive outcome.
Short-term changes in Symbol Digit Modalities Test (SDMT, oral version) | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The symbol Digit Modalities Test (SDMT) evaluates speeded information processing, perceptual and motor speed, and visual scanning. Higher scores indicate better cognitive outcome.
Short-term changes in Trail Making Test (TMT) | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The Trail Making Test (TMT) measures psychomotor speed and visual search attention (ie, visual scanning, graphomotor speed, and visuomotor processing speed), and executive functions (ie, working memory, inhibition control). TMT scores represent the time spent to complete the task and are provided in seconds. The higher the scores, the worse is the performance.
Short-term changes in Stroop Colour Word Test | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The Stroop Colour Word Test evaluates selective attention, cognitive flexibility and inhibition, and sensitivity to interference. Final score is obtained by computing the time interference effect (based on execution time) and the error interference effect (based on number of errors). Lower scores indicate better cognitive outcome.
Short-term changes in Frontal Assessment Battery (FAB) | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The Frontal Assessment Battery (FAB) evaluates executive functions (ie, conceptualization, verbal fluency, motor programming and executive control of action, self-regulation, resistance to interference, inhibitor control, environmental autonomy). Total scores range from 0 to 18. Higher scores indicate better cognitive outcome.
Short-term changes in Phonemic Verbal Fluency Test | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The Phonemic Verbal Fluency Test evaluate phonemic fluency by asking the patient to generate as many words as possible beginning with a specific letter. Higher scores indicate better cognitive outcome.
Short-term changes in EuroQoL-VAS (EQ-VAS) | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The EuroQoL-VAS (EQ-VAS) evaluates self-rated health on a vertical visual analogue scale (0: the worst health you can imagine; 100: the best health you can imagine). Higher scores indicate better health-related quality of life.
Short-term changes in Short Form Health Survey-12 (SF-12) | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The Short Form Survey-12 (SF-12) evaluates perceived physical health and mental health. Two subscores are generated, namely the physical component summary (PCS) and the mental component summary (MCS). Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Short-term changes in Generalized Anxiety Disorder-7 (GAD-7) | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The Generalized Anxiety Disorder-7 (GAD-7) evaluates anxiety symptoms severity in the last 2 weeks. Total scores range from 0 to 21. Higher scores indicate more severe anxiety.
Short-term changes in Patient Health Questionnaire-9 (PHQ-9) | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The Patient Health Questionnaire-9 (PHQ-9) evaluates depression symptoms severity in the last 2 weeks. Total scores range from 0 to 21. Higher scores indicate more severe depression.
Short-term changes in The Satisfaction-Profile (SAT-P) | From baseline (T0) to 4 weeks of rehabilitation (T1)
  The Satisfaction-Profile (SAT-P) evaluates patient's satisfaction with three different domains associated with HRQoL (ie, mood, resistance to physical fatigue, and mental efficiency) evaluated on a 10-cm horizontal visual analogue scale ranging from "extremely dissatisfied" to "extremely satisfied" (in the last month). Higher rates indicate higher patient's satisfaction.
Client-Centred Rehabilitation Questionnaire (CCRQ) | 4 weeks of rehabilitation (T1)
  The Client-Centred Rehabilitation Questionnaire (CCRQ) evaluates patient's subjective experience of care in rehabilitation settings (ie, patient participation in decision making and goal setting, patient-centred education, evaluation of outcomes from the patient's perspective, family involvement, emotional support, co-ordination/continuity, physical comfort). Total scores range from 33 to 165. Higher scores indicate better rehabilitation experience.
The Experience in Technology-based Rehabilitation Schedule (ExTR) | 4 weeks of rehabilitation (T1)
  The Experience in Technology-based Rehabilitation Schedule (ExTR) is an ad-hoc questionnaire measuring patients' experience of use of the devices. Specifically, technology learnability, acceptability, usefulness, adaptability, adverse effects, engagement, enjoyment, safety, and perceived effectiveness. Total scores range from 0 to 60. Higher scores indicate better patient's experience of use of the devices.
Psychosocial Impact of Assistive Device Scale (PIADS) | 4 weeks of rehabilitation (T1)
  The Psychosocial Impact of Assistive Device Scale (PIADS) evaluates the psychosocial impact of the technological devices. Each item is scored on a 7-point Likert scale. The score is meant to be either positive (+1, +2, +3 scores) or negative (-1, -2, -3 scores), with a central tendency marked as zero that indicates no perceived change after using the device. Higher scores reflect the technological device's stronger psychosocial impact
System Usability Scale (SUS) | 4 weeks of rehabilitation (T1)
  The System Usability Scale (SUS) evaluates perceived device usability (ie, devices ease-of-use and learnability). Total scores range from 0 to 100. Higher scores indicate higher usability.
Basic Activities of Daily Living (BADL) | 6-month telephone follow-up (T2)
  The Basic Activities of Daily Living (BADL) evaluates patient's level of independence in the basic activities in relation to the daily environment (ie, bathing, dressing, toilet, continence, transferring, feeding). Total scores range from 0 to 6. Higher scores indicate higher patient's autonomy.
Instrumental Activities of Daily Living (IADL) | 6-month telephone follow-up (T2)
  The Instrumental Activities of Daily Living (IADL) evaluates the patient's level of independence in performing more complex and instrumental activities (ie, using the telephone, making purchases, cooking, housekeeping, doing laundry, handling money, using means of transport, responsibility for his/her own medications). Total scores range from 0 to 8. Higher scores indicate higher patient's autonomy.
The telephone-based version of the MoCA (T-MoCA) | 6-month telephone follow-up (T2)
  The telephone-based version of the MoCA (T-MoCA) evaluates patient's global cognition (ie, attention, short-term and delayed verbal memory, language, and orientation to time and space). Total scores range from 0 to 15. Higher scores indicate better cognitive outcome.
Long-term changes in EuroQoL-VAS (EQ-VAS) | 6-month telephone follow-up (T2)
  The EuroQoL-VAS (EQ-VAS) evaluates self-rated health on a vertical visual analogue scale (0: the worst health you can imagine; 100: the best health you can imagine). Higher scores indicate better health-related quality of life.
Long-term changes in Short Form Health Survey-12 (SF-12) | 6-month telephone follow-up (T2)
  The Short Form Survey-12 (SF-12) evaluates perceived physical health and mental health. Two subscores are generated, namely the physical component summary (PCS) and the mental component summary (MCS). Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Patient Health Questionnaire-4 (PHQ-4) | 6-month telephone follow-up (T2)
  The Patient Health Questionnaire-4 (PHQ-4) evaluates patient's anxiety and depression symptoms severity in the last 2 weeks. Total scores range from 0 to 12. Higher scores indicate more severe anxiety and depression symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Pierobon, Dr., Principal Investigator — Istituti Clinici Scientifici Maugeri, IRCCS
Locations (1):
- Istituti Clinici Scientifici Maugeri, IRCCS, Pavia, PV, Italy

REFERENCES:
- [Derived] Zanatta F, Steca P, Fundaro C, Giardini A, Felicetti G, Panigazzi M, Arbasi G, Grilli C, D'Addario M, Pierobon A. Biopsychosocial effects and experience of use of robotic and virtual reality devices in neuromotor rehabilitation: A study protocol. PLoS One. 2023 Mar 10;18(3):e0282925. doi: 10.1371/journal.pone.0282925. eCollection 2023. PMID 36897863